CLINICAL TRIAL: NCT05344209
Title: A Randomized Phase II, Open-label, Multicenter Study Investigating Efficacy and Safety of Pembrolizumab +/- UV1 Vaccination as First Line Treatment in Patients With Inoperable Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Anti-PD-1/PD-L1 Treatment +/- UV1 Vaccination in Patients With Non-small Cell Lung Cancer
Acronym: LUNGVAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: University Hospital, Akershus (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); Helse Fonna (Other); Helse Nord-Trøndelag HF (Other); St. Olavs Hospital (Other); Alesund Hospital (Other); Helse Forde (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUNGVAC
Record Dates: First submitted 2022-03-30; First posted 2022-04-25 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Oncology; NSCLC Stage IV; NSCLC, Stage III
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Colony-Stimulating Factors; sargramostim

STUDY DESIGN:
Intervention Model Description: Randomized Phase II, Open-label, Multicenter Study
Masking Description: open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-PD-1/PD-L1 treatment + UV1 vaccination (Experimental): anti-PD-1/PD-L1 treatment + UV1 vaccination (and sagramostim)
  Interventions: Biological: UV1; Drug: Sagramostim; Drug: Anti-PD-1/PD-L1 treatment
- anti-PD-1/PD-L1 treatment (Other): anti-PD-1/PD-L1 treatment
  Interventions: Drug: Anti-PD-1/PD-L1 treatment

INTERVENTIONS:
Biological: UV1 — UV1 vaccine
  Arms: anti-PD-1/PD-L1 treatment + UV1 vaccination
Drug: Sagramostim — for stimulation of local dendritic cell population to take up the vaccine and to mature into professional APCs
  Other Names: leukine
  Arms: anti-PD-1/PD-L1 treatment + UV1 vaccination
Drug: Anti-PD-1/PD-L1 treatment — either pembrolizumab, atezolizumab or cemiplimab

SUMMARY:
A Randomized, Multicenter Study Investigating Efficacy and Safety of anti-PD-1/PD-L1-treatment +/- UV1 vaccination as first line treatment in patients with inoperable advanced or metastatic non-small cell lung cancer. The objective of the phase 2 study is to induce a meaningful Progression-Free Survival (PFS) benefit in patients with stage IIIB/IIIC or stage IV NSCLC by treating with anti-PD-1/PD-L1 treatment and UV1 vaccination versus anti-PD-1/PD-L1 treatment alone.

DETAILED DESCRIPTION:
The objective of the phase 2 study is to induce a meaningful Progression-Free Survival (PFS) benefit in patients with stage IIIB/IIIC or stage IV NSCLC by treating with anti-PD-1/PD-L1 treatment and UV1 vaccination versus anti-PD-1/PD-L1 treatment alone.

Patients are randomized to receive anti-PD-1/PD-L1 treatment until progression or unacceptable toxicity, for a maximum of 2 years, with or without 8 injections of 300 μg UV1 and 75 μg GM-CSF (UV1 vaccination). Patients randomized to UV1 vaccination, will start UV1 vaccination the same day as anti-PD-1/PD-L1 treatment is initiated, followed by three vaccinations over the next ten days. Thereafter, one vaccination per anti-PD-1/PD-L1 treatment cycle (c2-5), totaling to 8 UV1 vaccinations

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC stage IIIB/IIIC or IV not amenable for curative treatment, with PD-L1 ≥ 50% measured by a validated method, and eligible for pembrolizumab monotherapy in the first-line setting
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline according to RECIST 1.1
* Subjects who received previous neo-adjuvant or adjuvant systemic therapy (other than immunotherapies) will be eligible if neo-adjuvant or adjuvant therapy was completed at least 12 months prior to the development of metastatic disease. Last dose of neoadjuvant or adjuvant therapy must be more than 12 months prior to enrollment/randomization
* Available unstained archived tumour tissue sample in sufficient quantity to allow for analyses. At least fifteen unstained slides or a tumour block (preferred)
* Male and female age ≥ 18 years at time of signing the ICF
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ function as defined below
* Haemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
* Platelet count ≥100 x 109/L (>75,000 per mm3)
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL >40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min)

= Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

* Written informed consent obtained prior to any study specific procedure

Exclusion Criteria:

* Previous treatment with a PD-1 or PD-L1 inhibitor, including pembrolizumab or any other agent targeting immune checkpoints
* Previous malignancy (except non-melanoma skin cancer and the following in situ cancers: bladder, gastric, esophageal, colon, endometrial, cervical, melanoma or breast) unless a complete remission was achieved at least 2 years prior to study entry
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids (prednisone >10 mg or equivalent). Surgery, radiation and/or corticosteroids (any dose >10 mg prednisone equivalent) must have been completed ≥ 2 weeks prior to registration
* Known history of leptomeningeal carcinomatosis
* Uncontrolled seizures.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of pembrolizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroid premedication given as prophylaxis for imaging contrast allergy should not be counted for this criterion
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegner syndrome) within the past 2 years. Subjects with vitiligo, alopecia, Grave's disease, or psoriasis not requiring systemic treatment (within the past 3 years) are not excluded
* History of primary immunodeficiency
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Active infection including tuberculosis (clinical evaluation including: physical examination findings, radiographic findings, positive PPD test, etc.), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies as defined by a positive ELISA test). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. HIV testing is not required in the absence of clinical suspicion
* Pregnant or lactating women
* Live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving pembrolizumab
* Any condition that, in the opinion of the investigator, would interfere with the evaluation of study treatment or interpretation of patient safety or study results
* History of allergy or hypersensitivity to any of the active substances or excipients in the study drug
* Involvement in the planning and/or conduct of the study (investigator staff and/or staff at the study site)
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumours (RECIST 1.1) as determined by Blinded Independent Central Review (BICR) | Up to 2 years
  Evaluate and compare the efficacy of anti-PD-1/PD-L1-treatment with or without UV1 vaccination in patients with stage IIIB/IIIC or stage IV NSCLC.

SECONDARY OUTCOMES:
Response evaluation | Throughout trial (up to 2 years)
  Comparison of response rate according to RECIST v1.1 in patients who receive anti-PD-1/PD-L1 treatment and patients who receive anti-PD-1/PD-L1 treatment in combination with UV1.
monitoring AE | continously and until 4 months after discontinuation of study treatment
  evaluate safety and tolerability in patients who receive anti-PD-1/PD-L1 treatment and patients who receive anti-PD-1/PD-L1 treatment in combination with UV1.

OTHER OUTCOMES:
molecular characterization and analyses | up to 2 years
  investigate for possible biological markers for response, resistance and toxicity
immunophenotyping or characterization of the immune cell subsets in the periphery | In biological samples collected at screening, visit 5/6, end-of-treatment, safety visit and first follow-up visit.
  Investigate immunological responses.
To investigate the role of PET/CT in early response evaluation | up to 2 years
  PET-CT will be taken at predefined time-points for a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Odd Terje Brustugun, MD, PhD, Principal Investigator — Vestre Viken Health trust
Locations (1):
- Vestre Viken Health Trust, Drammen, Akershus, Norway